CLINICAL TRIAL: NCT01400776
Title: A Randomized, Double-Blind, Vehicle-Controlled Study of the Safety and Efficacy of WC3011 (Estradiol Vaginal Cream) in the Treatment of Symptoms of Vulvovaginal Atrophy in Postmenopausal Women
Brief Title: Safety & Efficacy WC3011 (Estradiol Vaginal Cream) in the Treatment of Vulvovaginal Atrophy in Postmenopausal Women
Acronym: VENUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-04409.3
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-09

CONDITIONS: Postmenopausal Vulvovaginal Atrophy
Keywords: Postmenopausal Women, Vaginal Dryness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- WC3011 Estradiol Vaginal Cream (2 Times/Week) (Experimental): WC3011 estradiol vaginal cream applied daily for 2 weeks, followed by dosing 2 times a week for 10 weeks.
  Interventions: Drug: WC3011 Estradiol Vaginal Cream
- Vehicle (2 Times/Week) (Placebo Comparator): Vehicle applied daily for 2 weeks, followed by dosing 2 times a week for 10 weeks.
  Interventions: Drug: Vehicle
- WC3011 Estradiol Vaginal Cream (3 Times/Week) (Experimental): WC3011 estradiol vaginal cream applied daily for 2 weeks, followed by dosing 3 times a week for 10 weeks.
  Interventions: Drug: WC3011 Estradiol Vaginal Cream
- Vehicle (3 Times/Week) (Placebo Comparator): Vehicle applied daily for 2 weeks, followed by dosing 3 times a week for 10 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: WC3011 Estradiol Vaginal Cream — WC3011 estradiol vaginal cream administered once daily for 2 weeks followed by 2X/week or 3X/week for 10 weeks, total treatment duration 12 weeks
  Arms: WC3011 Estradiol Vaginal Cream (2 Times/Week); WC3011 Estradiol Vaginal Cream (3 Times/Week)
Drug: Vehicle — Vehicle administered once daily for 2 weeks followed by 2X/week or 3X/week for 10 weeks, total treatment duration 12 weeks.
  Arms: Vehicle (2 Times/Week); Vehicle (3 Times/Week)

SUMMARY:
Study if WC3011 is effective and safe in the treatment of postmenopausal vaginal dryness due to vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females ≥35 years with either or both ovaries removed or naturally menopausal with moderate to severe vaginal dryness

Exclusion Criteria:

* Hypersensitivity to estrogen and/or progestin therapy
* Known or suspected premalignant or malignant disease (except successfully treated skin cancers)
* Manifestation of or treatment for significant cardiovascular disease, congestive heart failure, stroke or ischemic attacks
* Insulin-dependent diabetes mellitus
* Increased frequency or severity of headaches while on hormone or estrogen therapy
* Drug or alcohol addiction within last 2 years
* Participation in a clinical trial within 30 days
* Smoking ≥ 15 cigarettes daily
* Uncontrolled hypertension - systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥ 95 mmHg

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2012-02-27 (Actual); Study Completion 2012-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, PharmD, Study Director — Allergan
Locations (70):
- United States (70):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Mobile OB-GYN, PC, Mobile, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials, LLC, Phoenix, Arizona
  - Radiant Research-Scottsdale, Scottsdale, Arizona
  - Radiant Research-Tucson, Tucson, Arizona
  - Visions Clinical Research-tucson, Tucson, Arizona
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Healthcare Inc., San Diego, California
  - Physicians' Research Options LLC, Lakewood, Colorado
  - Costal Connecticut Resarch, LLC, New London, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - New Age Medical Research Corp, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - OB-GYN Specialists of the Palm, Palm Beach Gardens, Florida
  - Radiant Research-St. Petersburg, Pinellas Park, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Radiant Research-Atlanta, Atlanta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Atlanta North Gynecology, PC, Roswell, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Radiant Research-Chicago, Chicago, Illinois
  - Springfield Clinical, LLP, Springfield, Illinois
  - The South Bend Clinic, LLP, Granger, Indiana
  - Radiant Research - Overland Park, Overland Park, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Kentucky Pediatric Research, Inc., Bardstown, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - York Clinical Consulting, Marrero, Louisiana
  - Women Under Study, New Orleans, Louisiana
  - Beyer Research, Kalamazoo, Michigan
  - Ridgeview Research Two Twelve Medical Center, Chaska, Minnesota
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Lawrence OB-GYN Associates, P.C., Lawrenceville, New Jersey
  - Phoenix OB-GYN Assoc., LLC, Moorestown, New Jersey
  - The Center for Women's Health and Wellness, LLC, Plainsboro, New Jersey
  - Hawthorne Medical Research, Inc., Greensboro, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - The Columbus Center for Women's Health Research, Columbus, Ohio
  - HWC - Women's Research Center, Englewood, Ohio
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Advanced Clinical Research, Medford, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Susan L. Floyd, MD, PC, Wexford, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Practice Research Organization, Inc., Dallas, Texas
  - Radiant Research-Dallas, Dallas, Texas
  - Research Across America RHD Professional Plaza 4, Dallas, Texas
  - Advances in Health, Inc., Houston, Texas
  - Radiant Research-San Antonio, San Antonio, Texas
  - Center for Reproductive Medicine, Webster, Texas
  - J. Lewis Research-foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research - Foothill Family Clinic South, Salt Lake City, Utah
  - Physicians' Research Options LLC, Sandy City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Women's Center, Richmond, Virginia
  - Seattle Women's: Health, Research Gynecology, Seattle, Washington
  - North Spokane Women's Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Started | 238 | 124 | 237 | 123
Completed | 217 | 119 | 209 | 114
Not Completed | 21 | 5 | 28 | 9
Not completed — Adverse Event | 7 | 2 | 9 | 2
Not completed — Lost to Follow-up | 1 | 0 | 4 | 1
Not completed — Withdrew Consent | 4 | 2 | 6 | 1
Not completed — Protocol Deviation | 6 | 1 | 5 | 2
Not completed — Reason not Specified | 3 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week) | Total
Number analyzed (Participants) | 238 | 124 | 237 | 123 | 722
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (6.27) | 57.8 (6.34) | 58.0 (6.03) | 58.7 (6.58) | 58.2 (6.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 124 | 237 | 123 | 722
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 15 | 10 | 45
  Not Hispanic or Latino | 224 | 118 | 222 | 113 | 677
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 1 | 3
  Black or African American | 29 | 18 | 27 | 14 | 88
  White | 202 | 105 | 208 | 106 | 621
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant's Self-Assessment of Severity of Vaginal Dryness to Week 12/Final Visit
Description: The severity of vaginal dryness was assessed and recorded on a questionnaire by the participants using the following 4 point scale where, 0=None (The symptom is not present), 1=Mild (The symptom is present but may be intermittent; does not interfere with participants activities or lifestyle), 2=Moderate (The symptom is present. Participant is usually aware of the symptom, but activities and lifestyle are only occasionally affected), and 3=Severe (The symptom is present. Participant is usually aware and bothered by the symptom and have modified participant's activities and/or lifestyle due to the symptom. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12/Final Visit
Population: Modified Intent-to-Treat Population (mITT) included all participants in the safety population who had at least one postbaseline primary efficacy result. Number analyzed is the number of participants with evaluable data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 2.49 (0.50) | 2.46 (0.52) | 2.50 (0.50) | 2.50 (0.50)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 233 | 123 | 231 | 121
  Change from Baseline to Week 12/Final Visit | -1.27 (0.90) | -0.99 (0.89) | -1.31 (0.93) | -1.17 (0.97)

2. Primary Outcome: Change From Baseline in Vaginal pH to Week 12/Final Visit
Description: Vaginal pH was obtained at final visit of the study. The pH was a numeric value from a scale of 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12/Final Visit
Population: mITT Population included all participants in the safety population who had at least one postbaseline primary efficacy result. Number analyzed is the number of participants with evaluable data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 6.51 (0.96) | 6.49 (0.86) | 6.40 (0.93) | 6.40 (0.86)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 227 | 120 | 226 | 115
  Change from Baseline to Week 12/Final Visit | -1.08 (1.14) | -0.37 (0.92) | -0.99 (1.05) | -0.46 (0.90)

3. Primary Outcome: Change From Baseline in Percentage of Vaginal Superficial Cells to Week 12/Final Visit
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12/Final Visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 227 | 123 | 225 | 117
percentage of superficial cells
  Baseline | 0.85 (3.76) | 0.66 (1.62) | 0.79 (1.63) | 0.66 (1.21)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 205 | 114 | 202 | 104
  Change from Baseline to Week 12/Final Visit | 11.44 (14.74) | 3.05 (7.11) | 17.30 (19.27) | 4.02 (12.16)

4. Primary Outcome: Change From Baseline in Percentage of Vaginal Parabasal Cells to Week 12/Final Visit
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12/Final Visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 227 | 123 | 225 | 117
percentage of parabasal cells
  Baseline | 48.36 (43.46) | 47.78 (44.51) | 42.56 (41.03) | 45.24 (42.47)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 205 | 114 | 202 | 104
  Change from Baseline to Week 12/Final Visit | 41.7 (42.76) | -8.20 (29.56) | -38.5 (39.78) | -16.0 (32.75)

5. Secondary Outcome: Change From Baseline in Investigator's Assessment of Atrophy to Week 12 and Week 12/Final Visit
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to atrophy scored on a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 233 | 123 | 231 | 121
score on a scale
  Baseline | 1.88 (0.60) | 1.94 (0.70) | 1.90 (0.64) | 1.88 (0.63)
  Change from Baseline to Week 12: number analyzed (Participants) | 213 | 118 | 209 | 112
  Change from Baseline to Week 12 | -0.77 (0.80) | -0.47 (0.71) | -0.76 (0.81) | -0.44 (0.76)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 228 | 121 | 226 | 117
  Change from Baseline to Week 12/Final Visit | -0.74 (0.80) | -0.48 (0.72) | -0.75 (0.81) | -0.44 (0.77)

6. Secondary Outcome: Change From Baseline in Investigator's Assessment of Pallor to Week 12 and Week 12/Final Visit
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to pallor scored on a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 1.76 (0.67) | 1.72 (0.76) | 1.74 (0.70) | 1.83 (0.67)
  Change from Baseline to Week 12: number analyzed (Participants) | 213 | 118 | 209 | 112
  Change from Baseline to Week 12 | -0.73 (0.81) | -0.36 (0.75) | -0.78 (0.79) | -0.59 (0.81)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 228 | 121 | 226 | 117
  Change from Baseline to Week 12/Final Visit | -0.71 (0.82) | -0.39 (0.76) | -0.77 (0.80) | -0.59 (0.81)

7. Secondary Outcome: Change From Baseline in Investigator's Assessment of Vaginal Dryness to Week 12 and Week 12/Final Visit
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to vaginal dryness scored on a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 1.92 (0.68) | 1.85 (0.73) | 1.83 (0.75) | 1.87 (0.76)
  Change from Baseline to Week 12: number analyzed (Participants) | 213 | 118 | 209 | 112
  Change from Baseline to Week 12 | -0.94 (0.88) | -0.53 (0.82) | -0.90 (0.89) | -0.74 (0.91)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 228 | 121 | 226 | 117
  Change from Baseline to Week 12/Final Visit | -0.91 (0.89) | -0.55 (0.83) | -0.89 (0.90) | -0.76 (0.92)

8. Secondary Outcome: Change From Baseline in Investigator's Assessment of Friability to Week 12 and Week 12/Final Visit
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to friability scored on a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 1.04 (0.91) | 1.02 (0.94) | 0.94 (0.89) | 1.04 (0.93)
  Change from Baseline to Week 12: number analyzed (Participants) | 213 | 118 | 209 | 112
  Change from Baseline to Week 12 | -0.66 (0.90) | -0.47 (0.86) | -0.60 (0.87) | -0.52 (0.89)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 228 | 121 | 226 | 117
  Change from Baseline to Week 12/Final Visit | -0.64 (0.89) | -0.48 (0.86) | -0.61 (0.86) | -0.52 (0.89)

9. Secondary Outcome: Change From Baseline in Investigator's Assessment of Petechiae to Week 12 and Week 12/Final Visit
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to petechiae scored on a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Week 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 0.74 (0.78) | 0.89 (0.89) | 0.70 (0.83) | 0.71 (0.81)
  Change from Baseline to Week 12: number analyzed (Participants) | 213 | 118 | 209 | 112
  Change from Baseline to Week 12 | -0.47 (0.74) | -0.38 (0.72) | -0.47 (0.82) | -0.29 (0.73)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 228 | 121 | 226 | 117
  Change from Baseline to Week 12/Final Visit | -0.44 (0.73) | -0.40 (0.71) | -0.46 (0.82) | -0.30 (0.75)

10. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of Severity of Vaginal Dryness to Weeks 2, 4, 8 and 12
Description: Participant's self-assessment of symptoms of VVA (severity of vaginal dryness) was scored according to a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 2.49 (0.50) | 2.46 (0.52) | 2.50 (0.50) | 2.50 (0.50)
  Change from Baseline to Week 2: number analyzed (Participants) | 229 | 123 | 229 | 119
  Change from Baseline to Week 2 | -0.83 (0.86) | -0.79 (0.88) | -0.95 (0.90) | -0.79 (0.84)
  Change from Baseline to Week 4: number analyzed (Participants) | 227 | 123 | 227 | 120
  Change from Baseline to Week 4 | -1.07 (0.82) | -0.93 (0.90) | -1.12 (0.91) | -0.95 (0.90)
  Change from Baseline to Week 8: number analyzed (Participants) | 217 | 121 | 219 | 116
  Change from Baseline to Week 8 | -1.25 (0.84) | -1.02 (0.90) | -1.43 (0.90) | -1.11 (0.91)
  Change from Baseline to Week 12: number analyzed (Participants) | 216 | 119 | 209 | 113
  Change from Baseline to Week 12 | -1.30 (0.91) | -0.97 (0.90) | -1.36 (0.94) | -1.20 (0.98)

11. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of Vaginal and/or Vulvar Irritation/Itching to Weeks 2, 4, 8, 12 and Week 12/Final Visit
Description: Participant's self-assessment of symptoms of VVA (vaginal and/or vulvar irritation/itching) was scored according to a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 1.26 (0.96) | 1.33 (1.00) | 1.11 (0.96) | 1.20 (0.89)
  Change from Baseline to Week 2: number analyzed (Participants) | 229 | 123 | 229 | 119
  Change from Baseline to Week 2 | -0.54 (1.09) | -0.67 (0.95) | -0.48 (1.05) | -0.48 (1.04)
  Change from Baseline to Week 4: number analyzed (Participants) | 227 | 123 | 227 | 120
  Change from Baseline to Week 4 | -0.62 (1.14) | -0.71 (0.92) | -0.48 (1.08) | -0.65 (1.01)
  Change from Baseline to Week 8: number analyzed (Participants) | 217 | 121 | 219 | 116
  Change from Baseline to Week 8 | -0.71 (1.11) | -0.82 (1.03) | -0.57 (0.97) | -0.58 (1.00)
  Change from Baseline to Week 12: number analyzed (Participants) | 216 | 119 | 209 | 113
  Change from Baseline to Week 12 | -0.75 (1.03) | -0.74 (1.02) | -0.59 (1.04) | -0.70 (0.86)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 233 | 123 | 231 | 121
  Change from Baseline to Week 12/Final Visit | -0.74 (1.01) | -0.74 (1.03) | -0.58 (1.02) | -0.63 (0.92)

12. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of Dysuria (Painful or Difficult Urination) to Weeks 2, 4, 8, 12 and Week 12/Final Visit
Description: Participant's self-assessment of symptoms of VVA (dysuria) was scored according to a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 0.38 (0.70) | 0.49 (0.75) | 0.45 (0.75) | 0.53 (0.80)
  Change from Baseline to Week 2: number analyzed (Participants) | 229 | 123 | 229 | 119
  Change from Baseline to Week 2 | -0.24 (0.67) | -0.22 (0.71) | -0.28 (0.74) | -0.38 (0.77)
  Change from Baseline to Week 4: number analyzed (Participants) | 226 | 123 | 227 | 120
  Change from Baseline to Week 4 | -0.20 (0.68) | -0.30 (0.60) | -0.28 (0.76) | -0.42 (0.77)
  Change from Baseline to Week 8: number analyzed (Participants) | 217 | 121 | 219 | 116
  Change from Baseline to Week 8 | -0.20 (0.75) | -0.28 (0.72) | -0.32 (0.75) | -0.34 (0.85)
  Change from Baseline to Week 12: number analyzed (Participants) | 216 | 119 | 209 | 113
  Change from Baseline to Week 12 | -0.28 (0.68) | -0.28 (0.64) | -0.36 (0.72) | -0.41 (0.79)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 233 | 123 | 231 | 121
  Change from Baseline to Week 12/Final Visit | -0.27 (0.66) | -0.27 (0.64) | -0.34 (0.75) | -0.39 (0.78)

13. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of Dyspareunia (Pain Associated With Sexual Activity) to Weeks 2, 4, 8, 12 and Week 12/Final Visit
Description: Participant's self-assessment of symptoms of VVA (dyspareunia) was scored according to a 4-point scale where: 0= none, 1= mild, 2= moderate, or 3= severe. The negative change from Baseline indicates improvement. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 203 | 116 | 208 | 109
score on a scale
  Baseline | 2.29 (0.93) | 2.23 (0.88) | 2.29 (0.85) | 2.38 (0.86)
  Change from Baseline to Week 2: number analyzed (Participants) | 140 | 89 | 146 | 79
  Change from Baseline to Week 2 | -0.79 (1.06) | -0.78 (1.07) | -0.86 (1.06) | -0.67 (1.01)
  Change from Baseline to Week 4: number analyzed (Participants) | 138 | 86 | 151 | 78
  Change from Baseline to Week 4 | -1.04 (1.06) | -1.03 (0.90) | -1.06 (1.03) | -0.78 (0.91)
  Change from Baseline to Week 8: number analyzed (Participants) | 140 | 92 | 155 | 81
  Change from Baseline to Week 8 | -1.08 (1.01) | -1.04 (0.96) | -1.36 (0.97) | -1.07 (1.09)
  Change from Baseline to Week 12: number analyzed (Participants) | 141 | 86 | 153 | 76
  Change from Baseline to Week 12 | -1.15 (1.09) | -1.06 (0.96) | -1.39 (1.01) | -1.09 (1.05)
  Change from Baseline to Week 12/Final Visit: number analyzed (Participants) | 170 | 104 | 188 | 93
  Change from Baseline to Week 12/Final Visit | -1.15 (1.07) | -1.03 (1.00) | -1.35 (1.02) | -1.06 (1.07)

14. Secondary Outcome: Percentage of Participants With Vaginal Bleeding Associated With Sexual Activity as Per Participant's Self-Assessment to Weeks 2, 4, 8, 12 and Week 12/Final Visit
Description: Vaginal bleeding associated with sexual activity was assessed by participants as either "present" or "absent". Percentage of participants with assessment "present" are reported. Week 12/Final Visit is defined as the last available postbaseline assessment up to Week 12.
Time Frame: Baseline (Day 0) and Weeks 2, 4, 8, 12 and Week 12/Final visit
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
percentage of participants
  Baseline | 15.81 | 17.89 | 17.75 | 24.79
  Week 2: number analyzed (Participants) | 229 | 123 | 229 | 119
  Week 2 | 6.55 | 7.32 | 6.11 | 9.24
  Week 4: number analyzed (Participants) | 227 | 123 | 227 | 120
  Week 4 | 5.29 | 6.50 | 2.64 | 5.00
  Week 8: number analyzed (Participants) | 217 | 121 | 219 | 116
  Week 8 | 4.61 | 4.96 | 2.74 | 6.90
  Week 12: number analyzed (Participants) | 216 | 119 | 209 | 113
  Week 12 | 6.94 | 5.04 | 3.35 | 6.19
  Week 12/Final Visit: number analyzed (Participants) | 233 | 123 | 231 | 121
  Week 12/Final Visit | 6.44 | 4.88 | 3.03 | 5.79

15. Secondary Outcome: Change From Baseline in Vaginal pH to Week 12
Description: Vaginal pH was obtained at final visit of the study. The pH was a numeric value from a scale of 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 234 | 123 | 231 | 121
score on a scale
  Baseline | 6.51 (0.96) | 6.49 (0.86) | 6.40 (0.93) | 6.40 (0.86)
  Change from Baseline to Week 12: number analyzed (Participants) | 212 | 117 | 209 | 110
  Change from Baseline to Week 12 | -1.10 (1.15) | -0.34 (0.89) | -1.01 (1.06) | -0.47 (0.87)

16. Secondary Outcome: Change From Baseline in Percentage of Vaginal Superficial Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 227 | 123 | 225 | 117
percentage of superficial cells
  Baseline | 0.85 (3.76) | 0.66 (1.62) | 0.79 (1.63) | 0.66 (1.21)
  Change from Baseline to Week 12: number analyzed (Participants) | 191 | 111 | 183 | 100
  Change from Baseline to Week 12 | 11.66 (14.51) | 3.17 (7.02) | 17.66 (19.37) | 3.36 (10.31)

17. Secondary Outcome: Change From Baseline in Percentage of Vaginal Parabasal Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
Number analyzed (Participants) | 227 | 123 | 225 | 117
percentage of parabasal cells
  Baseline | 48.36 (43.46) | 47.78 (44.51) | 42.56 (41.03) | 45.24 (42.47)
  Change from Baseline to Week 12: number analyzed (Participants) | 191 | 111 | 183 | 100
  Change from Baseline to Week 12 | -42.3 (42.90) | -8.08 (29.90) | -39.5 (39.46) | -14.9 (31.93)

ADVERSE EVENTS:
Time Frame: From first dose through the last study visit (Up to 12 weeks)
Description: The safety population included all participants who were randomized and received at least one dose of study drug.
Arm/Group | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Vehicle (3 Times/Week)
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/124 | 0/237 | 0/123
Serious Adverse Events (participants affected / at risk) | 1/238 | 0/124 | 0/237 | 1/123
Other Adverse Events (participants affected / at risk) | 46/238 | 20/124 | 57/237 | 23/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WC3011 Estradiol Vaginal Cream (2 Times/Week) (N=238) | Vehicle (2 Times/Week) (N=124) | WC3011 Estradiol Vaginal Cream (3 Times/Week) (N=237) | Vehicle (3 Times/Week) (N=123)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WC3011 Estradiol Vaginal Cream (2 Times/Week) (N=238) | Vehicle (2 Times/Week) (N=124) | WC3011 Estradiol Vaginal Cream (3 Times/Week) (N=237) | Vehicle (3 Times/Week) (N=123)
Vulvovaginal mycotic infection (Infections and infestations) | 12 | 3 | 26 | 8
Vaginal discharge (Reproductive system and breast disorders) | 13 | 4 | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 5 | 12 | 2
Urinary tract infection (Infections and infestations) | 12 | 7 | 7 | 7
Nasopharyngitis (Infections and infestations) | 3 | 2 | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.